CLINICAL TRIAL: NCT05693428
Title: Changes in Blood Oxygen Transport Function and Body Energy Expenditure During Anaesthesia During Cardiac Surgery in Adults: a Randomized Clinical Trial
Brief Title: Influence of Anesthetics on Clinical Outcome During Cardiac Surgery in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Bekzat Baiterek, 2nd year doctoral student, anesthesiologist, resuscitator, Astana Medical University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2022-12-16; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: CHD - Coronary Heart Disease
Keywords: sevoflurane; isoflurane; propofol; Oxygen consumption; energy expenditure; oxygen transport; metabolic status
MeSH Terms: conditions — Coronary Artery Disease | interventions — Propofol; Isoflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (Other): Anesthesia
  Interventions: Drug: Propofol
- Isofluran (Other): Anesthesia
  Interventions: Drug: Isoflurane
- Sevofluran (Other): Anesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — To maintain anaesthesia in Group 1 P, propofol was used as an anaesthetic in a dose of 5-6 mg/kg/h intravenously on a perfusor.
  Other Names: Propofol;
  Arms: Propofol
Drug: Isoflurane — isoflurane was used as anaesthetice of - 1.1-1.2 MAC.
  Arms: Isofluran
Drug: Sevoflurane — sevoflurane was used as an anaesthetic in a dose of - 1.7-1.9 MAC
  Arms: Sevofluran

SUMMARY:
Abstract Cardiac surgery in adults is associated with the occurrence of post-operative complications. Even minor complications can increase the cost of their treatment. Given the potentially preventable nature of a number of these postoperative complications, preventive methods should be used to improve outcomes after cardiac surgery. One of them, is the choice of anaesthetic technique.

Objectives: To evaluate the effects of sevoflurane, isoflurane and propofol on blood oxygen transport function and body energy expenditure during cardiac surgery in adults.

Materials and methods. A total of 90 patients were included in the study. All patients were divided into 3 groups: 1- (n=30) included patients who were anesthetized with propofol. The second group (n=30) consisted of patients who underwent sevoflurane inhalation anaesthesia. Group 3 (n=30) was treated with isoflurane. All patients underwent coronary artery bypass grafting under cardiopulmonary bypass.

DETAILED DESCRIPTION:
Introduction Anaesthetic support for various types of cardiac surgery, such as coronary artery bypass grafting (CABG), heart valve repair or replacement, ascending aorta surgery, heart transplantation and surgical treatment of congenital heart disease, share many principles. Indirect calorimetry can be an indicator of homeostatic changes during surgery. Stress increases oxygen consumption (VO2) and during anaesthesia there is a decrease in VO2.

Cardiac surgery in adults is associated with the occurrence of postoperative complications [1]. Even minor complications, can increase the cost of their treatment. Given the potentially preventable nature of a number of these postoperative complications, preventive methods should be used to improve outcomes after cardiac surgery. One of them, is the choice of anaesthetic technique [2].

Tissues vary considerably in their sensitivity to hypoxia. Neurons tolerate hypoxia for only a few minutes, whereas the smooth muscles of the bladder go several days without oxygen. This has important implications for oxygen transport and monitoring of tissue hypoxia in patients. The mechanisms controlling the distribution of oxygen in the body are not fully understood (3). Increased oxygen extraction, the ratio of consumption to transport, has been associated with poor outcome after surgery. The authors note [4] a -65 ml decrease in oxygen consumption after general anaesthesia. Researchers [5,6] found that surgery and anaesthesia did not significantly affect oxygen consumption and energy expenditure during anaesthesia. However, Julia Jakobsson et al (2021) state that general anaesthesia reduced VO2 by approximately one third in elderly patients undergoing major abdominal surgery. These changes require further evaluation in relation to outcomes and surgery (7). Cerebral blood flow was reduced by 27.6% and cerebral vascular resistance by 51% at moderate propofol concentrations. Brain oxygen consumption was reduced by 18.2% [8]. Oxygen delivery (DO2) is an important marker of O2 transport than arterial blood oxygen saturation (SaO2). Anaesthetics (propofol or sevoflurane) had no significant effect on DO2 . In addition, no correlation was found between SaO2 and DO2. DO2 data may provide useful additional information about the patient's condition, especially with low SaO2 [9]. A decrease in metabolic rate during anaesthesia has been noted in patients with hypothermia, but this did not alter DO2. A significant decrease in O2ER might be partly due to a shift to the left of the oxyhemoglobin dissociation curve, as indicated by a decrease in P50 [10]. Oxygen consumption during general anaesthesia was independent of the type of anaesthetics. General anaesthesia leads to a marked decrease in oxygen consumption, but during recovery the O2 uptake can increase dramatically. Meperidine can suppress and reduce postoperative VO2 to the level observed after TIA [11]. Indirect calorimetry can be an indicator of homeostatic changes during surgery. Stress increases oxygen consumption and during anaesthesia there is a decrease in VO2 due to lack of kinetic energy as a cellular metabolic response to surgical trauma and anaesthesia. More research is needed to find out which oxygen consumption measurement system is the most appropriate for anaesthesia and what the VO2 limit values might be [12].

In view of the above opinion of the authors and the lack of studies that have shown the effects of sevoflurane, isoflurane and propofol on energy expenditure, blood oxygen and oxygen transport function, this needs to be further investigated.

Objectives: To evaluate the effects of sevoflurane, isoflurane and propofol on blood oxygen transport function and body energy expenditure during cardiac surgery in adults.

Methods Study type: single-centre prospective randomised clinical trial. The study includes data from 90 patients operated on at the Cardiosurgery Department of the RSE Medical Centre Hospital of the President's Affairs Administration of the Republic of Kazakhstan. All patients underwent coronary artery bypass grafting under cardiopulmonary bypass (CPB). This research work was conducted between 2021 and 2022. To calculate the sample size, we used the formula n=t2*D*N/confidence interval*N+t2*α, which will allow to identify the static significance of the study.

This research was approved by the Local bioethical committee of Non-commercial joint-stock company AMU №3 and written informed consent was obtained from all subjects.

All patients were divided into 3 groups: 1 (control group) (n=30) consisted of patients who underwent anaesthesia with propofol (P). The second group (n=30) were patients who received sevoflurane inhalation anaesthesia (S). Group 3 (n=30) with isoflurane (I).

The study was conducted in 5 stages:

1. determined the patient's baseline values before anaesthesia;
2. after tracheal intubation;
3. Before the CPB;
4. after the CPB;
5. The post-operative period. Before induction into anaesthesia, haemodynamic monitoring with Nihon Kohden monitors (Japan) was initiated on admission to the operating theatre. The right radial artery was catheterised for invasive systemic pressure monitoring and arterial blood sampling, then a catheter was inserted into the central jugular vein (under ultrasound machine control) and guided into the right atrium for mixed venous blood sampling.

Cardiac stroke volume was determined by transthoracic echocardiography (CS=end diastolic volume - end systolic volume). Cardiac output (CO=CS x heart rate), cardiac index (CI=CB/body surface area) were determined. Blood oxygen content was determined using the formula CaO2 (arterial blood gas ABG) and CvO2 (central mixed venous BG) = [(1.34 × Hb × SO2) + (PO2 × 0.031)] / 100, arteriovenous difference = CaO2-CvO2. Oxygen delivery was determined using the formula (DO2 = CI* CaO2), oxygen consumption (VO2 = Cardiac index (CI)*AVR or VO2 = CB × (CaO2 - CvO2) ~ CB × Hb × 1.34 × (SaO2 - SvO2) / 100).

In the second stage, after tracheal intubation, indirect calorimetry was used to determine VO2, energy expenditure during anaesthesia, using a "Spirometry" (Oxford, UK), which was connected to an endotracheal tube and continuously showed oxygen demand and energy expenditure. Additionally, cardiac output was determined using Fick's formula. In the third and fourth stages of anaesthesia the same tests (cardiac output, cardiac index, consumption, oxygen delivery and energy expenditure) were determined. In the last stage to assess the pharmaco-efficiency of anaesthetics, the consumption of muscle relaxants and opioid analgesics was calculated. The time of extubation and the time of transfer of the patient to the specialist department were determined.

All patients were given the same type of premedication: 30-40 minutes before surgery, 0.3 mg/kg promedol was administered intramuscularly. Patients continued to take their usual baseline drugs both before and on the day of surgery to prevent withdrawal syndrome and to reduce the risk of myocardial ischaemia in the perioperative period.

All patients in both groups were given fentanyl in a dose of 5-7 µg/kg, ketamine 1.5-2 mg/kg, and propofol 1-1.5 mg/kg intravenously fractionally. Pipecuronium bromide 0.04-0.07 mg/kg was used as muscle relaxant in all patients. To maintain anaesthesia in Group 1 P, propofol was used as an anaesthetic in a dose of 5-6 mg/kg/h intravenously on a perfusor (BBRAUN). In Group 2, sevoflurane was used as an anaesthetic in a dose of - 1.7-1.9 MAC. In Group 3 isoflurane was used as anaesthetic. In all groups fentanyl 100 µg intravenously was administered fractionally to increase heart rate and blood pressure, also pipecuronium bromide 2 mg intravenously for muscle relaxation. During CPB in all patients in all groups, propofol was used at a dose of 6 mg/kg/h intravenously via perfusion, analgesic regimen: fentanyl 100 µg intravenously every 30 min; myorelaxant piperonium bromide 2 mg every 40-60 min. Norepinephrine solution was administered at a dose of 0.05 µg/kg/min intravenously on perfusor after CPB in all patients at the same dosages in all groups.

Aim to use cardiotonic drugs:

1. in order to maintain mean arterial perfusion pressure (CPB causes cytokine storm and vasodilation).
2. for inotropic support (for reperfusion syndrome, resulting in a lower ejection fraction).

The depth of anaesthesia was monitored with a processed electroencephalogram, such as a BIS.

Statistical analysis was performed using IBM SPSS Statistics 20 package using one-factor analysis of variance for independent samples and nonparametric Kraskel Wallis test. The Kraskel-Wallis test was applied only to myorelaxant consumption, as the distribution was non-normal on this parameter. A Pearson and Spearman correlation analysis was also performed to determine the significance of the association between cardiac index and oxygen consumption, as well as energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* The age is over 40 years old.
* coronary revascularization or >50% stenosis on coronary angiography
* CHD. Multivessel coronary lesions.
* Participants of both sexes will be included in the study
* Signed informed consent

Exclusion Criteria:

* pregnancy (risk to the baby and the mother)
* allergenic patients (anaphylactic shock).
* vulnerable groups.
* current congestive heart failure;
* current unstable angina pectoris;
* preoperative hemodynamic instability, defined as the use of vasopressors;

Ages: 45 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Cardiac index | 1 year
  Cardiac stroke (CS) volume was determined by transthoracic echocardiography (CS =end diastolic volume-end systolic volume). Cardiac output (CO=CS x heart rate), cardiac index (CI=CO/body surface area) were determined.
Oxygen transport | 1 year
  Oxygen delivery was determined by the formula (DO2 = CI* CaO2)
Oxygen consumption | 1 year
  Oxygen consumption (VO2 = Cardiac index *AVD or VO2 = CO × (CaO2 - CvO2) ~ CB × Hb × 1,34 × (SaO2 - SvO2) / 100)
energy expenditure | 1 year
  energy expenditure during anaesthesia indirect calorimetry was used with the help of spirometry device "Spirometry" (UK Oxford) which was connected to the endotracheal tube and continuously showed oxygen demand and energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Alibek Kh Mustafin, Professor, Study Chair — Astana Medical University
Locations (1):
- Bekzat, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No